CLINICAL TRIAL: NCT05515159
Title: Blood Biomarkers in Electroconvulsive Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 51089
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Electroconvulsive Therapy; Depression; Blood Biomarkers
MeSH Terms: conditions — Depression | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECT group: patients undergoing electroconvulsive therapy for depression
  Interventions: Other: electroconvulsive therapy
- control group: healthy controls; patients undergoing electroconversion for atrial fibrillation

INTERVENTIONS:
Other: electroconvulsive therapy — electrical stimulation of the brain while the patient is under anesthesia.
  Groups: ECT group

SUMMARY:
The present multi-disciplinary study will assess blood biomarkers to investigate putative mechanisms of action of ECT. Laboratory findings will be correlated to clinical parameters, cognitive measures and psychometric outcome measures. The aim is to elucidate the underlying mechanisms for both treatment effects and cognitive side effects of ECT.

DETAILED DESCRIPTION:
Study hypothesis That a combined dataset of biomarker and clinical/ demographic data can be used to identify possible mechanisms of action for ECT or pathophysiological mechanisms underlying major depression.

The study is based on already (prospectively, observational) collected data and biological material:

* in the Regional ECT Register (Regionalt medisinsk kvalitetsregister for nevrostimulerende behandling i Helse Vest, Datatilsynets konsesjon 2012/5490),
* the ECT-MRI study approved by REK sørøst "2013/1032 ECT and neuroradiology" with its study specific biobank (Imdep)
* and the ECT biobank, (Forskningsbiobanken for nevrostimulerende behandling i Helse Vest (REK Vest 2017/925).

Biological samples and demographic/clinical data from those sources will be analyzed together.

All patients received the standard ECT treatment, as it is provided at the ECT-department at the Haukeland University Hospital.

Inclusion criteria:

Patients (age > 18) referred to the ECT-unit and accepted for treatment.

Exclusion criteria:

Patients unable to give informed consent

Data from the current study will be compared to data from the control groups in the ECT-MRI study:

1. a group of patients undergoing ECV for AF (controls 1) and
2. healthy controls undergoing the same investigations as the ECT patient group, but not receiving ECT or anesthesia (controls 2).

Clinical assessments Clinical assessments and monitoring was performed in accordance with the routine assessments at the section for ECT , Haukeland US and described in the Regional Register for ECT (Regionalt medisinsk kvalitetsregister for nevrostimulerende behandling i Helse Vest, Datatilsynets konsesjon 2012/5490).

Blood and saliva biomarkers We will analyze DNA, RNA and blood biomarkers that may be relevant for several hypotheses related to possible pathophysiological mechanisms of major depression, possible mechanisms of action of ECT and changes in biomarkers during depression treatment. Due to the constant progress in the field, the decision on which markers to analyze and how to perform the analyses should not be taken too early. However, candidate markers include neurotrophic factors (e.g. BDNF, CREB), neurotransmitters (e.g. GABA/Glutamate and relevant genetic markers), inflammation factors and markers of damage to the blood-brain barrier. Further, we will assess metabolomic changes from pre to post-treatment and other relevant blood biomarkers.

Genetic analysis (DNA, RNA), such as changes in RNA and DNA methylation from pre to posttreatment, might identify putative areas that are important for the biological mechanisms underlying ECT response and associated with depression /disease development. Further analyses might include Genome-wide association analyses of severe/ treatment resistant depression (GWAS) (patients vs healthy controls), Genome-wide association analyses of ECT response (responders vs nonresponders) and Epigenome-wide association (EWA) analyses of ECT response.

Studies so far suggest that effects of therapy of psychiatric disorders may be detected in peripheral blood. The information on methylation will be collected from both blood and saliva, and EWA analyses will also be performed on both. We will utilize longitudinal data to examine changes in methylation of ECT responders, non-responders and controls to establish possibly long-term and short-term epigenetic changes associated with ECT.

Metabolic and Proteomic analyses of ECT response In ongoing studies, we recently observed significant effects of ECT on serum tryptophan metabolites, including neuroprotective kynurenines. In this study, we will continue our analyses by increasing the sample size and expanding the number of metabolites and proteins that we will examine in relation to ECT response.

ELIGIBILITY:
Inclusion Criteria:

Patients (age > 18) referred to the ECT-unit and accepted for treatment.

Exclusion Criteria:

Patients unable to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (age > 18) referred to the ECT-unit and accepted for treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
change in levels of blood biomarkers | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on reasonable request